CLINICAL TRIAL: NCT05223894
Title: Epicardial Injection of Human Pluripotent Stem Cell-derived Cardiomyocytes to Treat Severe Chronic Heart Failure
Brief Title: Treating Heart Failure With hiPSC-CMs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Help Therapeutics (Industry)
Collaborators: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZMLiu
Record Dates: First submitted 2021-12-22; First posted 2022-02-04 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hiPSC-CM therapy (Experimental): Injection of allogenic human pluripotent stem cell-derived cardiomyocytes (hPSC-CMs) during coronary artery bypass grafting surgery. 100 million hPSC-CMs in 2.5-5 mL medium suspension will be injected into the myocardium.
  Interventions: Biological: hiPSC-CM therapy
- Control (Sham Comparator): Coronary artery bypass grafting surgery only.
  Interventions: Other: Control

INTERVENTIONS:
Biological: hiPSC-CM therapy — Injection of allogenic human pluripotent stem cell-derived cardiomyocytes (hPSC-CMs) during coronary artery bypass grafting surgery. 100 million hPSC-CMs in 2.5-5 mL medium suspension will be injected into the myocardium.
  Arms: hiPSC-CM therapy
Other: Control — Coronary artery bypass grafting surgery only.
  Arms: Control

SUMMARY:
Heart failure has a high morbidity and mortality because the heart is one of the least regenerative organs in the human body. Drug treatments for heart failure manage symptoms but do not restore lost myocytes. Cellular replacement therapy is a potential approach to repair damaged myocardial tissue, restore cardiac function, which has become a new strategy for the treatment of heart failure. The purpose of this study is to assess the safety and efficacy of intramyocardial delivery of cardiomyocytes at the time of coronary artery bypass grafting in patients with chronic heart failure.

DETAILED DESCRIPTION:
Patients with heart failure will be treated with allogenic human pluripotent stem cell-derived cardiomyocytes ( hPSC-CM ) from healthy donors. The cells will be injected directly into the myocardium at time of coronary artery bypass grafting. Patients will be assessed at 1, 3, 6 and 12 months after cell transplantation for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 35-75 (including 35 and 75).
2. Have signed the Informed Consent Form (ICF).
3. Patients have chronic left ventricular dysfunction.
4. Patients have NYHA Class III-IV cardiac function even after improved medication for the treatment of advanced chronic heart failure.
5. Patients have indications for Coronary Artery Bypass Grafting.
6. 20% ≤ LVEF ≤ 40% as determined by echocardiogram (data collected up to 3 months prior to inclusion evaluation are valid; data collected within 1 month since a myocardial infarction are invalid).
7. Weakening or absence of segmental regional wall motion as determined by standard imaging.

Exclusion Criteria:

1. PRA ≥ 20% or DSA-positive.
2. Patient received ICD transplantation, CRT or similar treatment.
3. Patients with valvular heart disease or received heart valvular disease
4. Patients received treatment of percutaneous transluminal coronary intervention (PCI)
5. Patients with atrial fibrillation
6. Patients previously suffered sustained ventricular tachycardia or sudden cardiac death.
7. Baseline glomerular filtration rate <30ml/min/1.73m2.
8. Liver dysfunction, as evidenced by enzymes (AST and ALT) greater than three times the ULN.
9. Hematological abnormality: A hematocrit <25% as determined by HCT, white blood cell<2500/ul or platelet values <100000/ul without another explanation.
10. Known, serious radiographic contrast allergy, penicillin allergy, streptomycin allergy.
11. Coagulopathy (INR>1.3) not due to a reversible cause.
12. Contra-indication to performance of a MRI scan.
13. Recipients of organ transplant.
14. Clinical history of malignancy within 5 years (patients with prior malignancy must be disease free for 5 years).
15. Non-cardiac condition that limits lifespan <1 year.
16. On chronic therapy with immunosuppressant medication, such as glucocorticoid and TNF-α antagonist.
17. Patients allergy to or cannot use immunosuppressant.
18. Serum positive for HIV, HBV, HCV, TP.
19. Currently enrolled other investigational therapeutic or device study.
20. Patients who are pregnant or breast feeding.
21. Other conditions that researchers consider not suitable to participate in this study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events(SAEs) within 1 month post-CABG surgery. | 1 Month Post-operation
  Incidence of serious adverse events(SAEs) within 1 month post-CABG surgery. These include death, fatal myocardial infarction, stroke, cardiac tamponade, cardiac perforation, hemodynamic ventricular arrhythmias (duration > 15s), and new allogeneic human neoplasms.

SECONDARY OUTCOMES:
Size of infracted myocardium assessed by MRI | Baseline, 1, 3, 6 and 12 Months Post-operation
  Size of infracted myocardium;
Left Ventricular systolic performance as assessed by MRI | Baseline, 1, 3, 6 and 12 Months Post-operation
  left ventricular side wall thickness at diastolic; interventricular septum thickness;
Left ventricular ejection fraction assessed by MRI | Baseline, 1, 3, 6 and 12 Months Post-operation
  left ventricular ejection fraction;
Overall Left Ventricular systolic performance as assessed by MRI | Baseline, 1, 3, 6 and 12 Months Post-operation
  left ventricular end-systolic volume and end-diastolic volume; stroke volume;
Cardiac output assessed by MRI | Baseline, 1, 3, 6 and 12 Months Post-operation
  cardiac output;
Myocardium density assessed by MRI | Baseline, 1, 3, 6 and 12 Months Post-operation
  myocardium density;
Left ventricular mass assessed by MRI | Baseline, 1, 3, 6 and 12 Months Post-operation
  left ventricular mass at diastolic;
Overall Left Ventricular systolic performance as assessed by Echocardiogram | Baseline, 1, 3, 6 and 12 Months Post-operation
  Interventricular septum thickness at diastolic; left ventricular posterior wall thickness at diastolic;
Left Ventricular systolic performance as assessed by Echocardiogram | Baseline, 1, 3, 6 and 12 Months Post-operation
  left ventricular end-systolic diameter and end-diastolic diameter; left atrial diameter;
Left ventricular ejection fraction assessed by Echocardiogram | Baseline, 1, 3, 6 and 12 Months Post-operation
  left ventricular ejection fraction;
Mitral flow pattern (E/A) assessed by Echocardiogram | Baseline, 1, 3, 6 and 12 Months Post-operation
  mitral flow pattern (E/A) ;
Overall Left Ventricular systolic performance as assessed by PET/ECT Scan | Baseline, 6 and 12 Months Post-operation
  Myocardium perfusion
Functional status by 6 minute walk test | Baseline, 1, 3, 6 and 12 Months Post-operation
  Evaluate Functional Capacity via the Six Minute Walk Test
Functional status by New York Heart Association (NYHA) Classification | Baseline, 1, 3, 6 and 12 Months Post-operation
  Evaluate Functional Capacity via New York Heart Association (NYHA) Class Determination.
  It classifies patients in one of four categories based on their limitations during physical activity; Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Minnesota Living With Heart Failure Questionnaire (MLHFQ) | Baseline, 1, 3, 6 and 12 Months Post-operation
  Evaluate Quality Of Life Changes via Minnesota Living with Heart Failure (MLHF). The Maximum possible scores being 105 and the minimum 0. Higher scores indicate a worse or worsening quality of life, while lower scores or decreasing scores indicate a better quality of life.
Incidence of Serious Adverse Events (SAE) | Baseline, 1~12Months Post-operation
  SAE justified (all undesirable or unintended diseases or laboratory and imaging disorders and symptoms that occur in subjects after CABG surgery and 12 months postoperative follow-up, or until the subject withdrawals from the study. AE grading will be based on Common Terminology Criteria for Adverse Events (CTCAE) V5.0.)
Incidence of severe arrhythmia | First month post-operatively
  Clinically significant arrhythmias will be recorded by Electrocardiogram monitoring
Changes in penal reactive antibodies (PRA) | Baseline, 1, 3, 6 and 12 Months Post-operation
  Changes in penal reactive antibodies (PRA) as assessed via blooddraw
Changes in donor specific antibodies (DSA) | Baseline, 1, 3, 6 and 12 Months Post-operation
  Changes in donor specific antibodies (DSA) as assessed via blooddraw
Changes in cytokines | Baseline,1, 3, 6 and 12 Months Post-operation
  Change in NT-proBNP as assessed via blooddraw

CONTACTS AND LOCATIONS:
Overall Officials: Zhongmin Liu, MD,phD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai east Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No